CLINICAL TRIAL: NCT03744429
Title: A Dietary Intervention to Modify Breast Milk Content in Obese Lactating Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 228407
Record Dates: First submitted 2018-10-31; First posted 2018-11-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2024-10

CONDITIONS: Effect of Diet on Breast Milk Composition
Keywords: Breast Milk; Mediterranean Diet
MeSH Terms: interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mediterranean Meal Plan (Experimental): This is a single arm study in which participants will receive meals that follow a Mediterranean diet plan for 4 weeks. Breast milk samples will be collected before, during, and after the intervention period.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Mediterranean Diet — Participants will be provided with meals that follow a Mediterranean meal plan.

SUMMARY:
This study is a nutrition research study designed to look at how healthy meals can influence the content of breast milk. Moms will be provided with meals that follow a Mediterranean diet pattern for 4 weeks. The goal of the study is to see if breast milk content changes over the 4 week period. The infants of the moms will also be included in the study to measure any changes in growth.

ELIGIBILITY:
Inclusion Criteria:

* ≤4.5 months postpartum
* BMI 30 - 50 kg/m2
* ≥ 18 years of age
* Singleton pregnancy
* Exclusive breastfeeding and plans to exclusively breastfeed for at least 6 months postpartum
* Mother has a breast pump
* Mother is willing to collect breast milk for a 24 hour period.

Exclusion Criteria:

* Pre-existing conditions (e.g. diabetes, hypertension, heart disease)
* Use of recreational drugs, tobacco, or alcohol
* Use of medications or supplements for which breastfeeding is contraindicated
* Child has internal metal which may be an NMR safety concern

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be breastfeeding.
Enrollment: 32 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in breast milk fat concentration by mid-infrared spectroscopy | The change in breast milk fat concentration will be assessed by mid-infrared spectroscopy by measuring the concentration before the participants begin the dietary intervention, 2 weeks into the intervention, and at the end of the 4-week intervention.
  The primary aim is to test whether the dietary intervention modifies the breast milk fat concentration of obese mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsey Fiecke, PhD, Principal Investigator — Arkansas Children's Nutrition Center
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided